CLINICAL TRIAL: NCT04219254
Title: A Phase 1/2a Clinical Trial of BI-1206, a Monoclonal Antibody to CD32b (FcγRIIB), in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Brief Title: A Study of BI-1206 in Combination With Pembrolizumab in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioInvent International AB (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-BI-1206-03
Record Dates: First submitted 2019-10-21; First posted 2020-01-07 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor, Adult
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Phase 1/2a, dose escalation, consecutive-cohort, open-label study trial of BI-1206 in combination with pembrolizumab
Masking Description: open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BI-1206 + Pembrolizumab 25mg/mL (MK-3475) (Experimental): BI-1206 administrated either IV or SC + Pembrolizumab 200mg administered IV every third week as a fixed dose will be used.
  Interventions: Drug: BI1206

INTERVENTIONS:
Drug: BI1206 — BI-1206 administrated either IV or SC every third week. Pembrolizumab 200mg administered IV every third week as a fixed dose will be used in Phase 1 and IIa.
  The mTPI2 Design will be used for both the IV and SC cohorts. ivRP2D and scRP2D to be used in Phase
  Other Names: Pembrolizumab 25mg/mL (MK-3475)

SUMMARY:
Phase 1/2a Clinical Trial of BI-1206, a Monoclonal Antibody to CD32b (FcγRIIB), in Combination with Pembrolizumab in Subjects with Advanced Solid Tumors

DETAILED DESCRIPTION:
This is a Phase 1/2a, multicenter, dose-finding, consecutive-cohort, open-label trial of BI-1206 in combination with pembrolizumab in subjects with advanced solid tumors.

The trial will consist of 2 main parts:

Phase 1 with 2 different sets of cohorts assessing IV or SC dosing, with dose escalation of BI-1206 and selection of the RP2D of IV dosing (ivRP2D) and the RP2D of SC dosing (scRP2D).

Phase 2a with 2 parts: a signal seeking and a dose optimization part. In the signal seeking part, subjects with uveal melanoma and Non-Small Cellular Lung Cancer (NSCLC) will be treated with Pembrolizumab intravenously and BI-1206 at the scRP2D subcutaneously. In the dose optimization part, subjects with NSCLC will be randomized into one of 3 expansion arms and treated with pembrolizumab and BI-1206 at the scRP2D.

Subjects will initially receive 3 cycles of therapy with pembrolizumab in combination with BI-1206, either IV or SC.

Subjects who show clinical benefit (CR, PR, or SD) at the Week 9 Visit may continue on combination therapy (pembrolizumab/BI-1206). Starting at Week 10, these subjects will receive additional cycles of pembrolizumab and BI-1206 every 3 weeks for up to 32 additional cycles or up to 2 years from their first dose of BI-1206 therapy or until progression.

Note: The study is only open for enrolling subjects into the phase 2a part.

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to provide written informed consent for the trial.
* Is ≥18 years of age on day of signing informed consent.
* Phase I only: Has a histologically confirmed advanced solid tumor. Subjects must have received at least 2 doses of an approved anti-PD-1/L1 mAb, and have documented progression on or within 12 weeks from the last dose of anti-PD-1/L1 mAb.
* For patients with NSCLC (phase 2A SC cohorts):

Have a histologically confirmed diagnosis of advanced or metastatic NSCLC and not have an EGFR sensitizing (activating) mutation or an ALK translocation.

Have a PD-L1 positive (TPS≥50%) tumor as determined by IHC at a local laboratory.

Have not received prior systemic immunotherapy or chemotherapy treatment for their advanced/metastatic NSCLC.

Have provided formalin-fixed tumor tissue sample from a biopsy of a tumor lesion either at the time of or after the diagnosis of advanced or metastatic disease has been made and from a lesion not previously irradiated to perform biomarker analysis.

• For patients with uveal melanoma (phase 2A SC cohort): Have a histologically confirmed diagnosis of advanced or metastatic uveal melanoma

Have a PD-L1 positive (TPS≥1%) tumor as determined by IHC at a local laboratory.

Have not received prior systemic immunotherapy or chemotherapy treatment for their advanced/metastatic uveal melanoma. Subjects who have received previous treatment with tebentafusp and/or liver directed therapy are allowed.

Have provided formalin-fixed tumor tissue sample from a biopsy of a tumor lesion either at the time of or after the diagnosis of advanced or metastatic disease has been made and from a site not previously irradiated to perform biomarker analysis.

* Phase I only: Is intolerant of, refuses, or is not eligible for standard antineoplastic therapy.
* Has at least 1 measurable disease lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
* Phase IIa only: Is willing to provide an archival tumor tissue sample or newly obtained [core, incisional, OR excisional] biopsy of a tumor lesion not previously irradiated.
* Is able to safely undergo a baseline tumor tissue biopsy prior to first dose of BI-1206.
* Has a life expectancy of ≥12 weeks.
* Has an ECOG performance status of 0-1.
* Has adequate organ function as confirmed by laboratory values listed in the main body of the protocol
* Phase IIa only: Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to enrolment
* Phase IIa only: Participants with history of HCV infection are eligible if HCV viral load is undetectable at Screening
* Phase IIa only: Has adequate hematological and biochemical indices as listed in the main body of the protocol

Exclusion Criteria:

* Needs doses of prednisolone >10 mg daily (or equipotent doses of other corticosteroids) while on the study, other than as premedication.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has known or suspected hypersensitivity to pembrolizumab or BI-1206 or any of their excipients.
* Has cardiac or renal amyloid light-chain (AL) amyloidosis.
* Has received radiotherapy within 2 weeks of the first dose of BI-1206.
* Has not recovered from AEs to at least Grade 1 by CTCAE v5.0 (or higher) due to prior anticancer therapies• Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active, known or suspected autoimmune disease.
* Is a female subject and has the ability to become pregnant (or already pregnant or lactating/breastfeeding)
* Is a male subject with partner(s) of childbearing potential (unless he agrees to use a barrier method of contraception during the study and for 12 months after completing treatment)
* Has had major surgery from which the subject has not yet recovered Is at high medical risk because of non-malignant systemic disease, including severe active infections on treatment with antibiotics, antifungals, or antivirals
* Has presence of chronic graft-versus-host disease.
* Has had an allogenic tissue/solid organ transplant.
* Has a known history of HIV infection
* Has a history of active tuberculosis (Bacillus tuberculosis)
* Has received a live vaccine within 30 days before the first dose of study treatment
* Has uncontrolled or significant cardiovascular disease as listed in the main body of the protocol
* Has a known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the study
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or lead to participation not being in the best interest of the subject, in the opinion of the treating Investigator.
* Is participating or planning to participate in another interventional clinical study or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study drug
* Has a known additional malignancy of another type, with the exception of adequately treated cone-biopsied carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) and basal or squamous cell carcinoma of the skin
* Has a diagnosis of primary or acquired immunodeficiency disorder or has taken any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Is unable to attend the study site to receive the study treatment

Additional exclusion criteria are described in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Estimated)
Dates: Start 2020-06-29 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Documentation of AEs and SAEs, clinically significant laboratory parameters, and physical findings, as well as their causality to BI-1206 and/or pembrolizumab administration | Up to 2 year
  Assess the safety and tolerability profile of increasing doses of BI-1206, administered IV or SC, in combination with pembrolizumab in subjects with advanced solid tumors
DLT occurrence; determination of signal-seeking dose, the MTD or maximum administered dose of BI-1206 in Phase 1, based on the mTPI-2 design | During the 42-day treatment period on induction therapy
  In Phase 1, identify DLTs, determine the MTD, and select a signal-seeking Phase 2a dose of BI-1206 given via IV infusion or SC injection in combination with pembrolizumab (administered at the standard dose of 200 mg every 3 weeks) to subjects with advanced solid tumors who are experiencing disease progression and have been previously treated with anti-PD-1 or anti- PD-L1 antibodies

SECONDARY OUTCOMES:
Determination of standard PK parameters (i.e., AUC, Cmax, Tmax, and terminal half-life [t½]) for BI-1206 | Up to 2 year
  Study the PK profile of BI-1206 administered IV or SC in combination with pembrolizumab in subjects with advanced solid tumors
Measurement of ADA response to BI-1206. | Up to 2 year
  Assess the immunogenicity of BI-1206, administered IV or SC, in subjects with advanced solid tumors, when given in combination with pembrolizumab.
Measurement of CD32b receptor occupancy on B cells. | Up to 2 year
  Evaluate the effect of BI-1206 IV or SC when administered in combination with pembrolizumab on CD32b receptor occupancy on B cells in subjects with advanced solid tumors.

OTHER OUTCOMES:
Assessment of best disease responses according to Immunological Response Evaluation Criteria in Solid Tumors (iRECIST). | 8 weeks after first dose BI1206 and every 9 weeks for subjects who continue on therapy
  Assess possible anti-tumor activity of BI-1206 administered IV or SC in combination with pembrolizumab, 8 weeks after first dose of BI-1206 (i.e., the Week 9 Visit), including follow-up confirmation for progressive disease (PD), in subjects with advanced solid tumors
Measurement of progression free survival. | Up to 2 year
  Assess the duration of clinical response to BI-1206 administered IV or SC in combination with pembrolizumab.
Measurement of duration of objective response and objective response rate | Up to 2 year
  Duration of response: Time-to-event estimates will be generated using the Kaplan-Meier method.
  Objective response rate: ORR is defined as the percentage of subjects who achieved CR or PR.
Measurement of peripheral blood B-lymphocyte counts | Up to 2 year
  Evaluate the effect of BI-1206 administered in combination with pembrolizumab on the depletion of peripheral blood B-lymphocytes in subjects with advanced solid tumors
Measurement of expression levels of immunological markers and/or other biomarkers in tissue biopsies and blood | Up to 2 year
  Study the expression levels of immunological markers and/or other biomarkers of cohort specific disease(s) and markers of treatment response in the tumor and/or peripheral blood and study the potential correlation of levels of expression with clinical responses
Measurement of BI-1206 and pembrolizumab presence in tissue biopsies using immunohistochemistry | Up to 2 year
  Evaluate the tumor penetrance of BI-1206 and pembrolizumab. Only applicable in Phase 1.
Determination of Fcγ receptor isoforms using nucleotide-based assays on genetic material extracted from whole blood and/or tissue | Up to 2 year
  Investigate the genetic background of participants with respect to FcγR isoforms and explore a potential correlation of the genetic background with clinical responses
Measurement of serum cytokine levels and/or soluble CD32b. | Up to 2 years
  Study the potential cause of infusion related reaction (IRR), such as cytokine release and/or soluble CD32b

CONTACTS AND LOCATIONS:
Locations (25):
- United States (5):
  - University of California Los Angeles, Los Angeles, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - HealthPartners Institute - Regions Cancer Care Center,, Saint Paul, Minnesota
  - Oklahoma University , Stephenson Cancer Center, Oklahoma City, Oklahoma
  - NEXT Oncology, San Antonio, Texas
- Georgia (3):
  - LTD High Technology Hospital Med Center, Batumi
  - Israel-Georgian Medical Research Clinic Helsicore, Tbilisi
  - Jerarsi Clinic, Tbilisi
- Germany (3):
  - Medizinische Hochschule Hannover, Hanover
  - Nationales Centrum für Tumorerkrankungen, Heidelberg
  - Universität des Saarlandes, Homburg
- Poland (3):
  - Maria Skłodowska-Curie National Institute of Oncology, Gliwice
  - Medical University of Silesia, Katowice
  - Instytut Centrum Zdrowia Matki Polki, Lodz
- Romania (2):
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta", Cluj-Napoca
  - Centrul de Oncologie SF Nectarie SRL, Craiova
- Spain (6):
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Universitari Vall D´Hebron, Barcelona
  - Institut Català d'Oncologia Hospital Duran i Reynals, Barcelona
  - Hospital Puerta de Hierro, Majadahonda
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Virgen de la Macarena, Seville
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Lund University Hospital, Lund
  - Karolinska University Hospital, Solna, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
All information concerning the product as well as any matter concerning the operation of the Sponsor, such as clinical indications for the drug, its formula, methods of manufacture and other scientific data relating to it, that have been provided by the Sponsor and are unpublished, are confidential and must remain the sole property of the Sponsor. The Investigator will agree to use the information only for the purposes of carrying out this studytrial and for no other purpose unless prior written permission from the Sponsor is obtained.
Supporting Information: Study Protocol
Time Frame: Within one year from end of study
Access Criteria: Paper copy of CSR